CLINICAL TRIAL: NCT02711891
Title: Topical Loperamide Gel for Pain Reduction During Repeat Finger Lancing: A Randomized Double Blind Trial
Brief Title: Topical Loperamide Gel for Pain Reduction During Repeat Finger Lancing
Acronym: Loperamide
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13091401-IRB02; IND 122919 (Other: Food and Drug Administration)
Record Dates: First submitted 2015-12-11; First posted 2016-03-17 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Pain
Keywords: fingerstick; opioid; heelstick; loperamide; topical opioid
MeSH Terms: conditions — Pain | interventions — Loperamide; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5% Loperamide gel (Experimental): Participants received 5% loperamide gel (0.2gm equivalent to 10 mg) applied following a single surgilance to the 5th digit. The loperamide gel was applied 10 minutes following the first lance, rubbed in for one minute within an 8 mm mold surrounding the lance site. The mold was removed and the gel was covered with a transparent occlusive dressing and left in place for 30 minutes. The forearm was also swabbed with the loperamide gel which was left in place for 30 minutes. The placebo gel contained the same ingredients without the loperamide. The loperamide gel formulation includes: Loperamide 5%, Propylene Glycol; Ethanol (190 proof USP); Ethyl acetate; and Klucel HF 1%.
  Interventions: Drug: Loperamide
- Placebo gel (Placebo Comparator): Participants received placebo gel (0.2gm) applied following a single surgilance to the 5th digit. The placebo gel was applied 10 minutes following the first lance, rubbed in for one minute within an 8 mm mold surrounding the lance site. The mold was removed and the gel was covered with a transparent occlusive dressing and left in place for 30 minutes. The forearm was also swabbed with the placebo gel which was left in place for 30 minutes. .The placebo gel contained the same ingredients without the loperamide. The placebo gel formulation includes: Propylene Glycol; Ethanol (190 proof USP); Ethyl acetate; and Klucel HF 1%.
  Interventions: Drug: Drug, placebo gel

INTERVENTIONS:
Drug: Loperamide — Following lance one, 0.2 grams of loperamide 5% gel was applied from a sterile syringe to the participants previous lance site within an 8 mm diameter circular plastic mold. The loperamide gel was rubbed lightly on the skin surface for one minute using a gloved finger swirled into the mold site. The mold was removed and the site was covered with a transparent occlusive dressing for 30 minutes. At 30 minutes the gel was removed with gauze, the skin cleaned with an alcohol wipe and the second lance was done within the same location as the first. The loperamide gel was also swabbed to the forearm within the 8 mm mold and left in place for 30 minutes.
  Arms: 5% Loperamide gel
Drug: Drug, placebo gel — Following lance one, 0.2 grams of gel alone was applied to the participants previous lance site within an 8mm diameter circular plastic mold. The gel was rubbed lightly on the skin surface for one minute using a gloved finger swirled into the mold site. The mold was removed and the site was covered with a transparent occlusive dressing left in place for 30 minutes. At 30 minutes the gel was removed with gauze, the skin cleaned with an alcohol wipe and the second lance was done within the same location as the first. The placebo gel was also swabbed to the forearm within the 8 mm mold and left in place for 30 minutes.
  Arms: Placebo gel

SUMMARY:
This study evaluates topical loperamide 5% gel in reducing pain during repeat finger lancing (finger stick) in healthy adults. Half of participants received 5% loperamide gel applied to their fingertip prior to their second lance and the other half received the gel only.

DETAILED DESCRIPTION:
Lancing the finger and heel to obtain capillary blood for specimen collection and diagnostic testing is a painful and tissue damaging procedure. With each lance, there is direct splicing of capillaries along with free nerve endings resulting in an immediate localized pain response and hyperalgesia from the release of pain producing substances. Opioid agonists (morphine, fentanyl, loperamide) have demonstrated significant analgesia when locally injected or topically applied to a site of inflammation/injury in animal models.

Loperamide, a piperdine derivative with a structure similar to the synthetic opioid meperidine, has strong affinity for Mu opioid receptors. It was approved by the FDA in 1969 as an anti-diarrheal agent with Mu opioid activity mimicked the constipating effects of other opioids, but with markedly reduced CNS effects due to its affinity for p-glycoprotein, preventing crossing the blood brain barrier (BBB) under normal circumstances.

This prospective, double-blind, repeated measures, randomized investigational new drug trial used loperamide developed as a topical gel in 34 adult participants to determine its analgesic effects during repeat finger lancing. The investigators also assessed for any local skin reaction to the gel application and for any constipation or abdominal cramping which might be evidence of systemic absorption and Mu opioid agonist activity on the gut.

This study would be applicable for use in 28.9 million adults who are diabetic and require finger lancing for blood glucose monitoring and the high risk newborn population who require repeat heel lancing for specimen collection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers willing to have 2 consecutive finger sticks completed.

Exclusion Criteria:

* Participants are excluded if they have a history of drug induced hypersensitivity reactions; took any anti-inflammatory medications in the past 12 hours; if they routinely performed finger lancing for blood specimen monitoring (e.g. diabetes); or had calloused fingers pads.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owens ME, Todt EH. Pain in infancy: neonatal reaction to a heel lance. Pain. 1984 Sep;20(1):77-86. doi: 10.1016/0304-3959(84)90813-3. PMID 6493791
- [Background] Fruhstorfer H, Schmelzeisen-Redeker G, Weiss T. Capillary blood volume and pain intensity depend on lancet penetration. Diabetes Care. 2000 Apr;23(4):562-3. doi: 10.2337/diacare.23.4.562. No abstract available. PMID 10857956
- [Background] Johnston CC, Strada ME. Acute pain response in infants: a multidimensional description. Pain. 1986 Mar;24(3):373-382. doi: 10.1016/0304-3959(86)90123-5. PMID 3960577
- [Background] Stein C. The control of pain in peripheral tissue by opioids. N Engl J Med. 1995 Jun 22;332(25):1685-90. doi: 10.1056/NEJM199506223322506. No abstract available. PMID 7760870
- [Background] Stein C, Schafer M, Machelska H. Attacking pain at its source: new perspectives on opioids. Nat Med. 2003 Aug;9(8):1003-8. doi: 10.1038/nm908. PMID 12894165
- [Background] DeHaven-Hudkins DL, Burgos LC, Cassel JA, Daubert JD, DeHaven RN, Mansson E, Nagasaka H, Yu G, Yaksh T. Loperamide (ADL 2-1294), an opioid antihyperalgesic agent with peripheral selectivity. J Pharmacol Exp Ther. 1999 Apr;289(1):494-502. PMID 10087042
- [Background] Nozaki-Taguchi N, Yaksh TL. Characterization of the antihyperalgesic action of a novel peripheral mu-opioid receptor agonist--loperamide. Anesthesiology. 1999 Jan;90(1):225-34. doi: 10.1097/00000542-199901000-00029. PMID 9915332
- [Background] Page GG. Are there long-term consequences of pain in newborn or very young infants? J Perinat Educ. 2004 Summer;13(3):10-7. doi: 10.1624/105812404X1725. PMID 17273395
- [Background] Osborne DW. (2002). Patent No. US 6355657 B1. US. https://www.google.com/patents/US6355657 Accessed June 1, 2014
- Available data/document: Study Protocol: Loperamide — http://www.rush.edu/clinical-trials-rush-university-medical-center — Contact the Rush Office of Research Affairs for all materials 312 942-5498
- Available data/document: Informed Consent Form: Loperamide — http://www.rush.edu/clinical-trials-rush-university-medical-center — Contact the Rush Office of Research Affairs for all materials 312 942-5498

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Individuals were excluded from participating if they had a history of drug induced hypersensitivity reactions; took any anti-inflammatory medications in the past 12 hours; if they routinely performed finger lancing for blood specimen monitoring (e.g. diabetes); or had calloused fingers pads.
Groups:
- 5% Loperamide Gel: Participants received 5% loperamide gel (0.2gm equivalent to 10 mg) applied following a single surgilance to the 5th digit. The loperamide gel was applied 10 minutes following the first lance, rubbed in for one minute within an 8 mm mold surrounding the lance site and then covered with a transparent occlusive dressing for 30 minutes. At 30 minutes the gel was removed with gauze, the skin cleaned with an alcohol wipe and the second lance was done within the same location as the first. The forearm was also swabbed with the loperamide gel which was left in place for 30 minutes. The loperamide gel formulation includes: Loperamide 5%, Propylene Glycol; Ethanol (190 proof USP); Ethyl acetate; and Klucel HF 1%.
Period: Overall Study
Arm/Group | 5% Loperamide Gel | Placebo Gel
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5% Loperamide Gel | Placebo Gel | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Full Range); unit: years] — The age range was 18-72 years and there was no difference in mean age between the loperamide group (M 42years) and the placebo group (M 39 years).
  years | 42 [18 to 72] | 39 [18 to 72] | 41.5 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34
Anxiety to needle stick scale [Mean (Standard Deviation); unit: units on a scale] — The anxiety about needle sticks scale range is 0-10 with 0 (0=not at all anxious) to 10 (worst imaginable). Prior to the first finger lance, participants were asked "How anxious (nervous) do you get about having a stick for blood drawing?" and circled their response on a print form as part of their demographic data.
  units on a scale | 2.8 (2.6) | 3.2 (2.6) | 2.9 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Pain - Numeric Rating Scale
Description: Subject responded to "Please mark the degree of pain you felt following the lance" and drew a line on a 0 (no pain) to 10 (worst possible pain) scale within one minute of the lance.
Time Frame: Within one minute following each lance
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pain Rating Loperamide Study Arm: The 5th digit finger pad of the non-dominant hand was cleaned with 70% alcohol. The participant was asked to look away and the finger pad was punctured using a single-use lancet which contains a stainless steel blade automatic trigger and retractor that incises with a 21 guage needle to a controlled depth of 2.2 mm and with of 0.8 mm. The pain rating was obtained within one minute following the lance. Ten minutes following lance one, 0.2 grams of Loperamide 5% gel was applied using a circular mold to the lance site and left in place for 30 minutes. At 30 minutes, the gel was removed, site cleansed with alcohol and lanced in the same location. The second pain rating was obtained within one minute of the lance.
- Pain Rating Placebo Study Arm: The 5th digit finger pad of the non-dominant hand was cleaned with 70% alcohol. The participant was asked to look away and the finger pad was punctured using a single-use lancet which contains a stainless steel blade automatic trigger and retractor that incises with a 21 guage needle to a controlled depth of 2.2 mm and with of 0.8 mm. The pain rating was obtained within one minute following the lance. Ten minutes following lance one, 0.2 grams of Placebo gel was applied using a circular mold to the lance site and left in place for 30 minutes. At 30 minutes, the gel was removed, site cleansed with alcohol and lanced in the same location. The second pain rating was obtained within one minute of the lance.
Arm/Group | Pain Rating Loperamide Study Arm | Pain Rating Placebo Study Arm
Number analyzed (Participants) | 17 | 17
units on a scale
  Basal Lance | 2.6 (1.7) | 2.5 (2.3)
  Lance 2 | 1.9 (1.4) | 4.2 (2.4)
Statistical Analysis 1: Comparison: Pain Rating Loperamide Study Arm; Test type: Superiority or Other; p = 0.8, Paired Sample T-test
Statistical Analysis 2: Comparison: Pain Rating Placebo Study Arm; Test type: Superiority or Other; p = .003, Paired Sample T-test
Statistical Analysis 3: Comparison: Pain Rating Loperamide Study Arm vs Pain Rating Placebo Study Arm; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

2. Primary Outcome: Pain - Comparative Pain Scale
Description: Within one minute following the second lance, subjects were asked "In comparison to the first finger stick, how would you rate the pain of the second": much less, a little less, about the same, a little more or much more.
Time Frame: Within one minute of the second lance, participants will be asked to circle their comparison pain rating to the first lance delivered 40 minutes earlier to the same digit.
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Loperamide Gel | Placebo Gel
Number analyzed (Participants) | 17 | 17
Participants
  Participants rating pain much less | 3 | 0
  Participants rating pain a little less | 5 | 0
  Participants rating pain a little more | 1 | 4
  Participants rating pain much more | 1 | 4
  Participants rating pain about the same | 7 | 9

3. Secondary Outcome: 24 Hour Numeric Pain (0 to 10 Scale) in the Lanced Finger Site.
Description: Numeric pain rating using the numeric rating scale 0-10 (0=no pain and 10 = worst pain ever) at 24 hours following finger lancing
Time Frame: 24 hours following the second lance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5% Loperamide Gel | Placebo Gel
Number analyzed (Participants) | 17 | 17
score on a scale | .23 (.56) | 1.23 (1.4)
Statistical Analysis 1: Comparison: 5% Loperamide Gel vs Placebo Gel; Test type: Superiority or Other; p = 0.01, t-test, 1 sided
Statistical Analysis 2: Comparison: 5% Loperamide Gel vs Placebo Gel; Test type: Superiority or Other; p = .001, Chi-squared

4. Secondary Outcome: 24 Hour Sensitivity in Lanced Finger to Touch and Pressure
Description: Sensitivity questions adapted from the pain quality assessment scale:
  After the application of the gel in both the treatment and control (Placebo) group, each participant from both groups was asked about the sensitivity of the fingerstick site to light or clothing rubbing against it over the past day (24 hours later), the sensitivity scale is as follows: (0=non-sensitive; 1-sensitive). A scale score of 0 means- a better outcome.
  After the application of the gel in both the treatment and control (Placebo) group, each participant from both groups was asked about the sensitivity of the fingerstick site when something was pressed against it over the past day (24 hours later), the sensitivity scale is as follows: (0=not tender and 1=tender). A scale score of 0 means- a better outcome.
Time Frame: 24 hours post lancing.
Population: 17 participants from both groups/arms were analyzed for this result outcome based on the score on the scale.
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Loperamide Gel | Placebo Gel
Number analyzed (Participants) | 17 | 17
Participants
  Proportion of participants with no sensitivity | 14 | 6
  Proportion with no sensitivity to pressure | 15 | 5

5. Secondary Outcome: Change in Beats Per Minute (BPM) Within Groups During Lance One and Lance Two Procedure
Description: BPM obtained using the Kenek Edge Pulse Oximeter System using a flipclop sensor and companion app. Mean BPM during lance initiation through recovery (30 seconds following lance) reported.
Time Frame: Average of BPM during each phase of the lance procedure (lance, specimen collection, recovery)
Population: Repeat measures lance one and lance two -
Measure: Mean (Standard Deviation); unit: beats per minute (Mean)
Groups:
- Loperamide Repeat Measure: For Loperamide group, BPM obtained using the Kenek Edge Pulse Oximeter System using a flipclop sensor and companion app. Mean BPM during lance initiation through recovery (30 seconds following lance) reported.
  Beat per minute average for each phase of the lance procedure.
- Placebo Repeat Measure: For Placebo group, BPM obtained using the Kenek Edge Pulse Oximeter System using a flipclop sensor and companion app. Mean BPM during lance initiation through recovery (30 seconds following lance) reported.
  Beat per minute average for each phase of the lance procedure.
Arm/Group | Loperamide Repeat Measure | Placebo Repeat Measure
Number analyzed (Participants) | 17 | 17
beats per minute (Mean)
  Lance One BPM Average | 74.6 (12.0) | 74.1 (9.4)
  Lance 2 BPM Average | 74.3 (11.4) | 71.8 (7.19)
Statistical Analysis 1: Comparison: Loperamide Repeat Measure vs Placebo Repeat Measure; The population BPM lance one = population BPM mean lance two. Loperamide 1= Loperamide 2. Placebo 1=Placebo 2; Test type: Superiority or Other; p = .876, t-test, 1 sided — Comparison of mean BPM during lance procedure for L1 vs L2 Loperamide
Statistical Analysis 2: Comparison: Loperamide Repeat Measure vs Placebo Repeat Measure; Mean HR during the procedure for lance one will equal mean HR lance two following loperamide gel applciation; Test type: Superiority or Other; p = .085, ANOVA — Comparison of the mean between HR one and HR two during the procedure for lance one will equal the mean HR lance two following loperamide gel application; df 16

6. Secondary Outcome: Safety- Number of Participants With Treatment Related Adverse Events as Assessed by the CTCAE V.4
Description: CTCAE will be utilized for reporting any adverse events with specific focus on skin and tissue disorders. A Standard erythema scale (0=no effect, 0.5=observer indecisive, 1=faint pink-no border, 1.5=faint pink border, 2=faint pink with one border, 2.5=fain pink with two borders, 3=red, 3.5=fiery red 4=violaceous red will also be used to classify skin erythema.
Time Frame: Direct observation of treatment site at one minute and 30 minutes. Participant report at 24 hours if any redness is present on the forearm.
Measure: Number; unit: participants
Arm/Group | 5% Loperamide Gel | Placebo Gel
Number analyzed (Participants) | 17 | 17
participants | 0 | 0

7. Secondary Outcome: Safety - Number of Participants With Treatment Related Adverse Gastrointestinal Disorders Using the CTCAE V. 4 With Focus on Abdominal Pain, Constipation and Diarrhea
Description: Participant report of any abdominal pain or change in stool pattern (constipation or diarrhea) over the past 24 hours using the CTCAE V.4 with focus on abdominal pain, constipation and diarrhea..
Time Frame: 24 hour participant report
Measure: Number; unit: participants
Arm/Group | 5% Loperamide Gel | Placebo Gel
Number analyzed (Participants) | 17 | 17
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected at 24 hours.
Arm/Group | 5% Loperamide Gel | Placebo Gel
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No